CLINICAL TRIAL: NCT03056807
Title: Evaluation of Apnea Tolerance in Bariatric Patients Following Rapid-sequence Induction of Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11506
Record Dates: First submitted 2017-01-30; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: General Surgery
Keywords: tolerable apneic time; bariatric surgery; gastric band surgery; intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person measuring and recording the study data ("timer") will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - 25° head-up position (Active Comparator): Participants will be positioned at a 25° head-up position for procedure.
  Interventions: Other: 25° head-up position
- B - 55° head-up position (Active Comparator): Participants will be positioned at a 55° head-up position for procedure.
  Interventions: Other: 55° head-up position

INTERVENTIONS:
Other: 25° head-up position — Angle person is positioned for procedure.
  Arms: A - 25° head-up position
Other: 55° head-up position — Angle person is positioned for procedure.
  Arms: B - 55° head-up position

SUMMARY:
The purpose of this study is to compare the effect of the 25° head-up position versus the 55° head-up position on tolerable apneic time (TAT) in bariatric patients scheduled for laparoscopic adjustable gastric band surgery following maximum preoxygenation and rapid-sequence induction (RSI) of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II-III patients
* Body Mass Index (BMI) of 40-60
* Scheduled for an elective laparoscopic adjustable gastric band surgery

Exclusion Criteria:

* Patients with abnormalities of the upper airway that require awake tracheal intubation
* Asthma
* Chronic obstructive pulmonary disease
* Pregnant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Tolerable Apneic Time (TAT) | Time between start of induction of general anesthesia (SpO2 100%) to decline of SpO2 94%, up to eight minutes
  Measure of the TAT between groups to determine if the TAT is a function of the participant's position.

SECONDARY OUTCOMES:
Length of time to intubation (TTI) | Time between start of the tracheal intubation procedure to completion of tracheal intubation, up to 2 minutes
Peripheral arterial hemoglobin oxygen saturation (SpO2) trough | Time until SpO2 decreased to 92%, up to 8 minutes
  Measure of the rebound SpO2. It is the lowest SpO2 reading reached subsequent to start of mechanical ventilation at the SpO2 value of 94% and it represents final completion of SpO2 decline.

CONTACTS AND LOCATIONS:
Overall Officials: Mirsad Dupanović, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States